CLINICAL TRIAL: NCT05909345
Title: Examination of Foot Posture's Change on Balance in Different Disorders
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: E-85646034-604.02.02-60261
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Back Pain; Knee Osteoarthritis
Keywords: back pain; Knee Osteoarthritis
MeSH Terms: conditions — Back Pain; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Knee Osteoarthritis
- Nonspecific Low Back Pain
- healthy peers

SUMMARY:
Foot; It is a terminal joint that opposes external resistance in the lower kinetic chain. It plays a primary role in weight transfer and ground response between the body and the ground.

DETAILED DESCRIPTION:
To investigate the extent to which foot posture affects balance and foot function in different disease groups. The amount of studies examining the effect of the postural structure of the foot and balance seen in different disease groups in the literature is insufficient.

ELIGIBILITY:
Inclusion criteria;

* Being between the ages of 45 - 65,
* Volunteer. Exclusion criteria;
* Having a musculoskeletal or neuromuscular disease that limits mobility,
* Presence of lower extremity sequelae,

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To evaluate the foot postures and balances of individuals with knee osteoarthritis and nonspecific low back pain.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Navicular Drop Test | one day
  The distance between the tubercle of the navicular, which is the attachment of the tibialis posterior muscle, and the ground, was measured in this position by asking each participant to give full weight to their bare feet. The distance between the navicular tubercle and the ground was measured without any weight on the feet in the subtalar neutral position. The difference between this distance and the amount of navicular height was recorded as navicular drop (millimetres).
Foot Posture Index | one day
  Foot Posture consists of palpation of 6 regions. Each criterion is evaluated between -2 and +2 and this result is noted. Positive values indicate pronation, negative values indicate supination.
Y Balance Test | one day
  The leg lengths of all individuals are measured bilaterally. While measuring, individuals are asked to lie in their anterior, posteromedial and posterolateral directions. Each of the participants is informed before the measurement. Measurements were made in both legs and will be repeated 3 times. When calculating the total score, the values in centimeters of the 3 directions are added. Divide by the product of the length of the leg by 3 and multiply the result by 100 to reach the percentile.

SECONDARY OUTCOMES:
Oswestry Low Back Pain Disability Questionnaire | one day
  It includes 1 item about pain and 9 items about activities of daily living. Each item is measured on a 6-point rank scale between 0 and 5 points according to the scenarios it contains. At the end of the survey, scores are summed up and a high score means loss of disability.
Western Ontario and MacMaster (WOMAC) | one day
  Western Ontario and MacMaster (WOMAC) is evaluated by dividing it into three groups as pain, stiffness and physical function, consisting of a total of 24 questions used in the evaluation of lower extremity OA. The total WOMAC score is obtained by summing up all the values by evaluating these three titles separately. At the end of the questionnaire, scores are summed up and a high score means loss of disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol hospital, Istanbul, Istanbul Avrupa Kitasi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sporndly-Nees S, Dasberg B, Nielsen RO, Boesen MI, Langberg H. The navicular position test - a reliable measure of the navicular bone position during rest and loading. Int J Sports Phys Ther. 2011 Sep;6(3):199-205. PMID 21904698